CLINICAL TRIAL: NCT02960880
Title: Real-world Comparative Effectiveness of Stroke Prevention in Patients With Atrial Fibrillation Treated With Rivaroxaban vs. Vitamin k Antagonists
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 18735
Record Dates: First submitted 2016-10-12; First posted 2016-11-10 (Estimated); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Atrial Fibrillation
Keywords: Rivaroxaban, Phenprocoumon, retrospective cohort study, Non-Valvular Atrial fibrillation, NVAF
MeSH Terms: conditions — Atrial Fibrillation | interventions — Rivaroxaban; Phenprocoumon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Rivaroxaban: NVAF patients who were newly initiated on Rivaroxaban for stroke prevention
  Interventions: Drug: Rivaroxaban (Xarelto, BAY597939)
- Phenprocoumon: NVAF patients who were newly initiated on Phenprocoumon for stroke prevention
  Interventions: Drug: Phenprocoumon (branded and generics)

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY597939) — 15mg, 20mg
  Groups: Rivaroxaban
Drug: Phenprocoumon (branded and generics) — Individually adjusted dose
  Groups: Phenprocoumon

SUMMARY:
The aim of this study is to assess the real world comparative effectiveness of Rivaroxaban prescribed in non-valvular atrial fibrillation (NVAF) routine care patients in Germany.

ELIGIBILITY:
Inclusion Criteria:

* First dispense date of Rivaroxaban (15mg or 20mg - PZN based) or Phenprocoumon (PZN based) between January 1, 2012 and December 31, 2015
* At least two verified outpatient diagnoses or one inpatient diagnosis (main or secondary diagnosis) of NVAF (ICD-10 GM I48.0/I48.1/I48.2/I48.9) in the individual time frame of 4 quarters before the index date (pre-index period) or within the index quarter
* Patients will be required to have 4 quarters of enrollment for the assessment of baseline characteristics and be observable and insured in the database for at least one day after their individual index date (post-index period)
* ≥ 18 years of age

Exclusion Criteria:

* Patients with valvular AF [4 quarters prior to the index date]
* Pregnancy [4 quarters prior to index date]
* Malignant cancers [4 quarters prior to the index date or "condition after"]
* Transient cause of AF [4 quarters prior to index date]
* Patients with VTE (pulmonary embolism or DVT) [60 days before index]
* Patients with major surgery defined as hip or knee replacement [60 days before index]
* Prescriptions of OACs (Rivaroxaban, VKA, Dabigatran, Apixaban) before index date [4 quarters prior to index date]
* Patients receiving more than one anticoagulant substance (Apixaban, Dabigatran, Rivaroxaban or Phenprocoumon) or more than one dosage of a substance on the index date
* For sensitivity analysis : Patient with any of the events defined in the combined endpoints [4 quarters prior to index date or "condition after"
* Patients with dialysis [4 quarters prior to index date]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients newly initiated with Rivaroxaban or Phenprocoumon with an NVAF diagnosis from January 1, 2012 through December 31, 2015. Patients will be identified from the HRI research database, a complete longitudinal dataset of patients under statutory health insurance in Germany.
Sampling Method: Non-Probability Sample
Enrollment: 99999 (Actual)
Dates: Start 2016-10-15 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Risk of ischemic stroke estimated as the number of hospitalizations with the ICD-10-GM diagnosis | Within time of drug exposure (Retrospective period of 5 years and 3 months)
Risk of intracranial hemorrhage (ICH) estimated as the number of hospitalizations with the ICD-10-GM diagnosis | Within time of drug exposure (Retrospective period of 5 years and 3 months)

SECONDARY OUTCOMES:
Risk of ischemic stroke or ICH estimated as the number of hospitalizations with the respective ICD-10-GM diagnosis | Within time of drug exposure (Retrospective period of 5 years and 3 months)
Risk of systemic embolism (SE) estimated as the number of hospitalizations with the ICD-10-GM diagnosis | Within time of drug exposure (Retrospective period of 5 years and 3 months)
Risk of transient ischemic attack (TIA) estimated as the number of hospitalizations with the ICD-10-GM diagnosis | Within time of drug exposure (Retrospective period of 5 years and 3 months)
Risk of ischemic stroke or SE or TIA estimated as the number of hospitalizations with the respective ICD-10-GM diagnosis | Within time of drug exposure (Retrospective period of 5 years and 3 months)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, Germany